CLINICAL TRIAL: NCT01728116
Title: A Randomized, Multi-Center, Pivotal Efficacy and Safety Study Comparing the EndoBarrier Gastrointestinal Liner System vs. Sham for Glycemic Improvement in Inadequately Controlled Obese Type 2 Diabetic Subjects on Oral Anti-Diabetes Agents
Brief Title: Safety and Efficacy of EndoBarrier in Subjects With Type 2 Diabetes Who Are Obese
Acronym: ENDO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Higher than anticipated rate of Hepatic abscess (N=7)
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-1
Record Dates: First submitted 2012-11-13; First posted 2012-11-16 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: glycemic control, type 2 diabetes, device, obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device (EndoBarrier) (Experimental): Device for glycemic control
  Interventions: Device: EndoBarrier
- Sham Procedure (Sham Comparator): sham procedure
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: EndoBarrier — Endoscopically-delivered and removable device comprised of an anchor that is placed in the duodenal bulb and a 60 cm long impermeable liner that passes distal from the anchor point
  Other Names: Duodenal-jejunal bypass liner (DJBL)
  Arms: Device (EndoBarrier)
Procedure: Sham Procedure — Endoscopic evaluation but no device placement
  Arms: Sham Procedure

SUMMARY:
To determine if the EndoBarrier safely and effectively improves glycemic control in obese subjects with type 2 diabetes

DETAILED DESCRIPTION:
This is a randomized, double blinded, prospective study. Subjects will be evaluated and randomized to either the device or sham treatment group if they qualify for the study. A comparison of glycemic control between the two groups will be assessed as the primary outcome measurement as well as the safety profile of the device.

ELIGIBILITY:
Inclusion Criteria:

* Males/females aged ≥ 21 years and ≤ 65 years
* Diagnosis of Type 2 Diabetes for ≤ 20 years
* Obese individuals (BMI ≥ 30 kg/m2 and ≤ 55 kg/m2)
* Stable doses (at least 3 months) of up to two anti-T2DM medications (MET, SU, DPP-4i or TZD)
* Glycemic state: HbA1c at screening ≥ 7.5% and ≤ 10.0%.
* Subjects willing to comply with study requirements
* Subjects who have signed an informed consent form

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus or having any history of ketoacidosis
* C-peptide < 1.0 ng/mL
* Triglyceride level > 400 mg/dL
* Vitamin D deficiency (<20 ng/mL)
* Male subjects with serum Creatinine >1.5 mg/dl or female subjects with Creatinine >1.4 mg/dL
* Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/microliter, or known coagulopathy
* Height < 5 feet (152.4 cm)
* Current alcohol or drug addiction
* Symptomatic kidney stones or gallstones within 6 months prior to randomization
* Chronic pancreatitis or acute pancreatitis within 12 months of randomization
* Diagnosis of osteoporosis or currently taking bisphosphonates or teriparatide
* Diagnosis of an autoimmune connective tissue disorder (e.g., lupus erythematosus, scleroderma)
* Active gastroesophageal reflux disease [GERD] uncontrolled with a Proton Pump Inhibitor (PPI)
* Thyroid disease unless controlled with medication
* Currently taking Non-Steroidal Anti-Inflammatory Drugs [NSAIDs] (e.g., aspirin, ibuprofen, etc.) within 10 days prior to randomization and/or there is a need or expected use of these agents during the trial 12 months post index procedure
* Currently taking prescription antithrombotic therapy (e.g., anticoagulant or antiplatelet agent) within 10 days prior to randomization and/or there is a need or expected need to use during the trial 12 months post index procedure
* Currently taking systemic corticosteroids, drugs known to affect GI motility, prescription/over-the-counter weight loss medications, or medications known to cause significant weight gain or weight loss within 30 days prior to randomization and/or there is a need or expected need to use these medications during the trial 12 months post index procedure
* Medication for type 2 diabetes other than MET, SU, DPP-4i, and TZD (e.g., GLP1 or insulin) within 3 months of screening
* Chronic use of narcotics, opiates, benzodiazepines, or other addictive tranquilizers
* Allergy or hypersensitivity to ceftriaxone, cephalosporins, penicillin, or any equivalent antibiotics
* Active Helicobacter pylori infection (Note: Subjects may be eligible after undergoing 2 weeks of antibiotic treatment without re-screening)
* Previous GI surgery or abnormal GI anatomical finding that could preclude the ability to place the EndoBarrier device, liner or affect the function of the liner
* Abnormal pathologies or conditions of the gastrointestinal tract, including current ulcers or Crohn's disease, history of atresias or untreated stenoses, current upper gastrointestinal bleeding conditions within 3 months of randomization
* Any condition or major illness that places the subject at undue risk by participating in the study
* Poor dentition not allowing complete chewing of food
* Enrolled in another investigational study within 3 months of screening for this study (Enrollment in observational studies is permitted)
* Residing in a location without ready access to study site medical resources
* Documented weight loss of >10 pounds anytime during the 3 months preceding randomization
* Positive stool guaiac at time of screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2012-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Kaplan, MD, PhD, Study Chair — Massachusetts General Hospital; Keith Gersin, MD, Study Director — Carolinas Medical Center
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Little Rock Diagnostic Center (LRDC), Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado/ Anschutz Health & Wellness Center, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Kentucky Research Group, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Beth Israel Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Legacy Research Institute, Portland, Oregon
  - Endocrinology Consultants of East Tennessee & Gastrointestinal Associates, Knoxville, Tennessee
  - Dallas Diabetes, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: GI Dynamics website — http://www.gidynamics.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 500 subjects were planned to be randomized into either the EndoBarrier or the sham control arm at a 2:1 ratio, respectively. Due to early termination of the trial, only 325 subjects were randomized with 216 EndoBarrier subjects and 109 sham control subjects.
Pre-assignment Details: The mITT population for the primary analyses includes 213 EndoBarrier subjects and 107 sham control subjects. The remaining five (5) subjects (n=3 randomized to device; n=2 randomized to sham) were deemed ineligible before an attempted device placement due to findings identified during the upper endoscopy.
Groups:
- EndoBarrier Group: Subjects randomized to the device group received the EndoBarrier Gastrointestinal Liner. Subjects also received a prophylactic dose of antibiotics on Procedure Day. Fluoroscopy was also used in conjunction with endoscopy to aid implantation of the EndoBarrier device. Medical Nutritional Therapy (MNT) counseling (as defined by the 2012 American Diabetes Association guidelines) was to be conducted at Baseline then Weeks 13, 26, 39, and 52 for both groups, and additionally at Week 65 for the EndoBarrier group.
- Sham Control Group: Subjects randomized to the sham control group also underwent an upper endoscopy (without fluoroscopy) according to standard institutional endoscopy practices. Subjects also received a prophylactic dose of antibiotics on Procedure Day.Medical Nutritional Therapy (MNT) counseling (as defined by the 2012 American Diabetes Association guidelines) was to be conducted at Baseline then Weeks 13, 26, 39, and 52.
Period: Overall Study
Arm/Group | EndoBarrier Group | Sham Control Group
Started | 213 (EndoBarrier mITT Subjects) | 107 (Sham mITT subjects)
Completed | 52 (Completed to Week 78) | 60 (Completed to Week 52)
Not Completed | 161 | 47
Not completed — Sponsor Terminated Study | 106 | 35
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Adverse Event | 13 | 0
Not completed — Procedure/device failure | 7 | 0
Not completed — Lost to Follow-up | 9 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Subject Non-Compliance | 2 | 0
Not completed — Inter-current finding at procedure | 1 | 0
Not completed — Incorrectly enrolled in Study | 0 | 1
Not completed — various not noted previously | 5 | 0

BASELINE CHARACTERISTICS:
Population: mITT
Groups:
- EndoBarrier Group: Subjects randomized to the device group received the EndoBarrier Gastrointestinal Liner. Subjects also received a prophylactic dose of antibiotics on Procedure Day. Fluoroscopy was also used in conjunction with endoscopy to aid implantation of the EndoBarrier device.
- Sham Control Group: Subjects randomized to the sham control group also underwent an upper endoscopy (without fluoroscopy) according to standard institutional endoscopy practices. Subjects also received a prophylactic dose of antibiotics on Procedure Day.
- Total: Total of all reporting groups
Arm/Group | EndoBarrier Group | Sham Control Group | Total
Number analyzed (Participants) | 213 | 107 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, range 25 to 65 years
  years | 52.9 (8.19) | 51.8 (8.21) | 52.5 (8.20)
Gender [Count of Participants; unit: Participants] — In both arms (Device and Sham) of the mITT population, 61.3% were female and 38.8% were male
  Participants
    Female | 127 | 69 | 196
    Male | 86 | 38 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 14 | 33
  Not Hispanic or Latino | 194 | 93 | 287
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Subjects were allowed to select more than one race.
  participants
    American Indian or Alaska Native | 6 | 3 | 9
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 44 | 22 | 66
    White | 165 | 80 | 245
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 1 | 1 | 2
Baseline Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 245.0 (47.46) | 245.6 (44.20) | 245.2 (46.32)
Baseline BMI [Mean (Standard Deviation); unit: kg/m2] | 38.4 (5.74) | 38.3 (5.33) | 38.4 (5.60)
HbA1c (%) fasting bloodwork [Mean (Standard Deviation); unit: percent] | 8.8 (0.92) | 8.9 (0.89) | 8.8 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Improvement in HbA1c
Description: Mean Change in HbA1c from Baseline to 12 Months in the mITT population with Bayesian Imputation
Time Frame: Baseline and12 months
Population: All randomized subjects who at their baseline endoscopy are judged to be potential recipients of the device (meaning no abnormal pathologies and/or conditions are present). Any subject who has a device enter their body, regardless of eligibility or randomization assignment, is also included in the treatment arm of the mITT population.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 213 | 107
Percentage of HbA1c | -1.07 (1.5) | -0.31 (1.59)

2. Primary Outcome: Primary Safety Endpoint: Early Device Removal Due to Device-Related SAE
Description: Of the 161 subjects for whom data were available at 12 Months, 19 (11.8%) subjects experienced device-related SAEs that required an early device removal.
Time Frame: Baseline and 12 Months
Population: mITT without Imputation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EndoBarrier Group
Number analyzed (Participants) | 161
percentage of participants | 11.8 [7.8 to 17.7]

3. Secondary Outcome: Assessment of Total Cholesterol Change at 12 Months Compared to Baseline
Time Frame: Baseline and 12 Months
Population: mITT population without imputation
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- EndoBarrier Group: Subjects randomized to the device group received the EndoBarrier Gastrointestinal Liner. MITT population without imputation
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 135 | 61
mg/dL | -11.30 (34.39) | -4.16 (47.14)

4. Secondary Outcome: Percentage of Subjects Who Achieve HbA1c Less Than or Equal to 7.0% at 12 Months
Time Frame: Baseline and 12 Months
Population: mITT population without imputation
Measure: Number; unit: percentage of participants
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 135 | 61
percentage of participants | 34.81 | 9.84

5. Secondary Outcome: LDL Change From Baseline
Time Frame: Baseline and 12 Months
Population: mITT without imputation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 133 | 59
mg/dL | -10.76 (31.42) | -10.54 (40.35)

6. Secondary Outcome: Triglycerides Change From Baseline
Time Frame: Baseline and 12 Months
Population: mITT population without imputation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 135 | 61
mg/dL | -41.50 (105.76) | 2.26 (96.04)

7. Secondary Outcome: Fasting Glucose Change From Baseline
Time Frame: Baseline and 12 Months
Population: mITT population without imputation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 135 | 61
mg/dL | -38.90 (66.08) | 5.31 (73.65)

8. Secondary Outcome: Systolic BP Change From Baseline
Time Frame: Baseline and 12 Months
Population: mITT population without imputation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 134 | 59
mmHg | -2.76 (17.07) | 1.22 (16.47)

9. Secondary Outcome: Diastolic BP Change From Baseline
Time Frame: Baseline and 12 Months
Population: mITT population without imputation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 134 | 59
mmHg | -2.02 (9.91) | 1.51 (11.19)

10. Secondary Outcome: Percentage of Subjects Who Achieve % Total Body Weight Loss Greater Than or Equal to 5% at 12 Months
Time Frame: Baseline and 12 Months
Population: mITT population without imputation
Measure: Number; unit: percentage of participants
Arm/Group | EndoBarrier Group | Sham Control Group
Number analyzed (Participants) | 135 | 60
percentage of participants | 60.74 | 20.00

ADVERSE EVENTS:
Time Frame: 18 months for device subjects, 12 months for sham subjects
Description: The calculation of SAE rates uses the denominator of 212 for the EndoBarrier group; this is the number of subjects who had a device implant attempted (i.e., passed through the mouth of the subject regardless of a successful implant or not).
Arm/Group | EndoBarrier Group | Sham Control Group
Serious Adverse Events (participants affected / at risk) | 53/212 | 5/108
Other Adverse Events (participants affected / at risk) | 206/212 | 96/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier Group (N=212) | Sham Control Group (N=108)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 8 (9) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Adhesion (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Complication of device removal (General disorders) | 1 (1) | 0 (0)
Obstruction (General disorders) | 4 (4) | 0 (0)
Pseudopolyp (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Esophageal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier Group (N=212) | Sham Control Group (N=108)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 1 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Corneal lesion (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 3 (3) | 1 (1)
Visual impairment (Eye disorders) | 3 (3) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 75 (96) | 14 (17)
Abdominal distension (Gastrointestinal disorders) | 45 (55) | 13 (13)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 125 (223) | 22 (29)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 7 (7) | 3 (4)
Barrett's oesophagus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Bezoar (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 57 (62) | 14 (16)
Diarrhoea (Gastrointestinal disorders) | 57 (74) | 39 (49)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 9 (9) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 15 (17) | 3 (3)
Faecal incontinence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 29 (33) | 6 (6)
Frequent bowel movements (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (18) | 9 (9)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 111 (164) | 24 (27)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 3 (5) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 2 (3) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 68 (85) | 9 (9)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 7 (7) | 0 (0)
Chest discomfort (General disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 5 (5) | 1 (1)
Device dislocation (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 27 (28) | 8 (9)
Feeling cold (General disorders) | 1 (1) | 2 (2)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 1 (1)
Obstruction (General disorders) | 2 (2) | 0 (0)
Oedema mucosal (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (4)
Pseudopolyp (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 10 (13) | 4 (5)
Temperature intolerance (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 9 (9) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 9 (9) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (3)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 3 (3) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (5) | 5 (7)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 2 (2)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 3 (3) | 2 (3)
Gingival infection (Infections and infestations) | 1 (3) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (4) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 10 (10) | 5 (5)
Nasopharyngitis (Infections and infestations) | 20 (20) | 13 (16)
Pneumonia (Infections and infestations) | 6 (6) | 3 (3)
Respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 6 (8) | 5 (5)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 2 (2)
Trichomoniasis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 16 (17) | 7 (7)
Urinary tract infection (Infections and infestations) | 9 (10) | 2 (2)
Vaginitis bacterial (Infections and infestations) | 2 (2) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 2 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Oesophageal injury (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Amylase decreased (Investigations) | 3 (4) | 0 (0)
Blood albumin abnormal (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 5 (6) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 2 (2) | 1 (1)
Blood chloride decreased (Investigations) | 3 (3) | 0 (0)
Blood cholesterol decreased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 6 (6) | 2 (2)
Blood creatinine decreased (Investigations) | 3 (4) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Blood electrolytes decreased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 3 (3) | 2 (2)
Blood iron decreased (Investigations) | 24 (27) | 9 (10)
Blood iron increased (Investigations) | 1 (2) | 0 (0)
Blood magnesium decreased (Investigations) | 9 (9) | 7 (7)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 4 (4) | 2 (2)
Blood triglycerides increased (Investigations) | 5 (5) | 4 (4)
Blood urea increased (Investigations) | 1 (1) | 3 (3)
Carbon dioxide decreased (Investigations) | 1 (1) | 2 (2)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 8 (10) | 8 (9)
Haematocrit decreased (Investigations) | 3 (4) | 3 (3)
Haematocrit increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 6 (7) | 1 (1)
Haemoglobin increased (Investigations) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (2) | 0 (0)
High density lipoprotein decreased (Investigations) | 2 (2) | 0 (0)
Insulin C-peptide increased (Investigations) | 1 (1) | 0 (0)
Iron binding capacity total increased (Investigations) | 4 (4) | 2 (2)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Lipase decreased (Investigations) | 5 (5) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lipids increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein decreased (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 4 (4) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (2) | 1 (1)
QRS axis abnormal (Investigations) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 3 (5) | 1 (1)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Transferrin saturation decreased (Investigations) | 21 (28) | 13 (16)
Transferrin saturation increased (Investigations) | 1 (1) | 0 (0)
Vitamin B12 decreased (Investigations) | 11 (13) | 1 (1)
Vitamin B12 increased (Investigations) | 2 (2) | 1 (1)
Vitamin D decreased (Investigations) | 14 (15) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 3 (8) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 36 (72) | 12 (33)
Hyperuricaemia (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 42 (45) | 14 (14)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 14 (14) | 12 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 45 (56) | 9 (9)
Bone loss (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 11 (12) | 3 (4)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 24 (25) | 18 (23)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Poor quality sleep (Nervous system disorders) | 2 (2) | 0 (0)
Sciatic nerve neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Fallopian tube disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 40 (54) | 22 (25)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Artificial crown procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Rhinoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic disorder (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 3 (4) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The ENDO Trial was stopped early due to a higher than anticipated rate of hepatic abscess (n=7).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI to provide to Sponsor for review at least sixty (60) days in advance of submission for publication. Sponsor reserves the right to delete any Confidential Information or other proprietary information of Sponsor (including trade secrets but not including Results) from the proposed publication or presentation.